CLINICAL TRIAL: NCT06128811
Title: The Use of DryShield and Rubber Dam Isolation Systems Among Pediatric Patients With Different Airway Patency: A Randomized Clinical Trial
Brief Title: Dental Isolation Systems Among Pediatric Patients With Different Airway Patency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Sara M.Bagher, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 134-11-22
Record Dates: First submitted 2023-11-01; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Airway Obstruction; Pain; Behavior
MeSH Terms: conditions — Airway Obstruction; Pain; Behavior | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: It is a split-mouth randomized clinical trial. And both sides fissure sealants will be provided at the same appointment by the same trained and calibrated dentist
Who Masked: Investigator
Masking Description: The statistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants who will receive rubber dam isolation followed by DryShieled will be considered group 1.
  Interventions: Device: Rubber Dam Isolation; Device: DryShieled isolation; Other: fissure sealant
- Group 2 (Active Comparator): Participants who will receive DryShieled followed by rubber dam isolation will be considered group 2.
  Interventions: Device: Rubber Dam Isolation; Device: DryShieled isolation; Other: fissure sealant

INTERVENTIONS:
Device: Rubber Dam Isolation — Rubber dam isolation will be placed using a proper size dental clamp on the first permanent molar after topical anesthesia application.
Device: DryShieled isolation — For the DryShieled isolation, a pedo-size mouthpiece will be utilized with all the participants.
Other: fissure sealant — After proper isolation, fissure sealant (Conseal-F TM SDI) will be applied following the manufacturer's instructions, and the quality of the applied fissure sealant will be checked with an explorer. An additional layer will be applied if any deficiency is detected

SUMMARY:
This randomized clinical trial will aim to evaluate the effect of DryShield isolation (DSI) and Rubber Dam isolation (RDI) systems on arterial oxygen saturation (SpO2), heart rate (HR), blood pressure (BP), behavior, subjective pain and discomfort, and time required among children with different airway patency based on Modified Mallampati classification (MMC). Healthy, cooperative 6-12-year-old children who need fissure sealant in at least two contralateral fully erupted permanent first molars will be included. The airway patency will be determined using MMC by two trained and calibrated dentists. Participants will be categorized based on their MMC score into patent airway (MMC Class I and II) and non-patent airway (MMC Class III and IV). During the treatment, the dental procedure will be videotaped, and the vital signs, including SpO2, HR, and BP, will be recorded every three minutes. A Validated Arabic Version of the Wong-Baker Pain Rating and the Face, Legs, Activity, Cry, Consolability (FLACC) scales will be utilized to record the participants' pain levels. In contrast, Frankl's Behavior will record their behavior during the dental procedure. Following the dental treatment, the participants' subjective pain and discomfort will be evaluated using a previously validated Arabic interview questionnaire.

DETAILED DESCRIPTION:
This study will aim to evaluate the effect of DryShield isolation system and rubber dam isolation on arterial oxygen saturation, heart rate, blood pressure, behavior, subjective pain and discomfort, and time required among 6-12-years-old healthy children with different airway patency based on Modified Mallampati classification scores.

This split-mouth randomized clinical trial will be conducted in the Pediatric Dentistry Department at King Abdulaziz University Dental Hospital Faculty of Dentistry (KAUDH) after obtaining ethical approval from the Research Ethics Committee at King Abdulaziz University.

Healthy, cooperative 6-12-year-old children who need fissure sealants in at least two contralateral fully erupted permanent first molars will be included. Children with partially erupted, previously restored, or carious first molars, children with uncooperative behavior during their previous dental treatment, children with fixed orthodontic appliances, and children with nasal obstruction will be excluded.

Children attending the pediatric dentistry clinics during the study period will be screened for eligibility. The parents or guardians of eligible children will be approached and given information about the study, including the risks, benefits, and drawbacks. If they agree to participate, an Arabic consent and assent form will be signed, and a treatment appointment will be scheduled. The airway patency assessment will be performed during the screening visit by two trained and calibrated dentists using Modified Mallampati classification scores. The participants will be asked to sit upright with their chin parallel to the floor, open their mouths to the maximum, and protrude their tongue without phonation to determine their Modified Mallampati classification score, ranging from one to four. Class I indicates that the soft palate, fauces, uvula, and tonsillar pillars are clearly visible. Class II means the soft palate, fauces, and the uvula are visible, while Class III is when only the soft palate and base of the uvula are visible. Finally, Class IV is when the soft palate is not visible. (13) Participants will be categorized based on their Modified Mallampati classification scores into two groups: patent airway (Class I and II) and non-patent airway (Class III and IV).

If a participant has more than two contralateral and fully erupted permanent first molars, only one pair of molars will be randomly selected to be included in the study.

At the scheduled appointment, the participants' age, sex, and previous experience with dental isolation will be recorded. Five minutes after the participant is seated on the dental chair, a pulse oximeter (OxyWatch, ChoiceMMed, Hamburg, Germany) will be placed on the right forefinger to record the SpO2 and HR as a baseline, and an automatic BP cuff will be applied to the left upper to record the baseline BP. The SpO2, HR, and BP will be recorded at three-minute intervals until the removal of the isolation system. Additionally, a stopwatch will measure the chair time required to complete the entire dental procedure. The time needed to assemble the RDI or the DSI will not be included. Also, only topical anesthesia will be applied before RD clamp application.

Both fissure sealants will be provided at the same appointment by the same trained and calibrated dentist. The Tell-Show-Do behavior management technique will be utilized with all participants. The dental procedure will be videotaped using a high-resolution camera fixed in the clinic. The recorded videos will be used to assess the participants' behavioral pain and discomfort using the Face, Legs, Activity, Cry, Consolability (FLACC) scale and behavior using Frankl behavior classification by two trained and calibrated evaluators independently.

For the DSI, a pedo-size mouthpiece will be utilized with all the participants. After proper isolation, fissure sealant (Conseal-F TM SDI) will be applied following the manufacturer's instructions.

After the fissure sealant procedure, the participants' subjective pain and discomfort will be evaluated using a validated Arabic Version of the Wong-Baker Pain Rating Scale and a previously validated Arabic interview questionnaire. The questionnaire will ask the participants to rate their experience on a numerical scale from zero to 10, with zero meaning "no irritating factor at all" and 10 indicating "presence of irritating factor all the time." The factors included noise, gagging sensation, fluid leak, stretching, pressure, pain, and discomfort associated with the isolation system.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy
2. Cooperative
3. 6-12-year-old children
4. Who need fissure sealants in at least two contralateral fully erupted permanent first molar

Exclusion Criteria:

1. Children with partially erupted, previously restored, or carious first molars.
2. Children with uncooperative behavior during their previous dental treatment.
3. Children with fixed orthodontic appliances
4. Children with nasal obstruction

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygen saturation | Baseline before starting the dental procedure and then during the procedure at three-minute intervals until the removal of the isolation system.
  Five minutes after the participant is seated on the dental chair, a pulse oximeter (OxyWatch, ChoiceMMed, Hamburg, Germany) will be placed on the right forefinger to record the arterial oxygen saturation.
Behavior | During the dental procedure.
  The dental procedure will be videotaped using a high-resolution camera fixed in the clinic. The recorded videos will be used to assess the participants's behavior using Frankl behavior classification by two trained and calibrated evaluators independently.
Subjective pain and discomfort | immediately after the end of the dental procedure.
  The participants' subjective pain and discomfort will be evaluated using a validated Arabic Version of the Wong-Baker Pain Rating Scale and a previously validated Arabic interview questionnaire.
Time required in minutes | During the dental procedure.
  A stopwatch will be used to measure the chair-time required to complete the entire dental procedure in minutes.
Heart rate per minute (beat per minute) | Baseline before starting the dental procedure and then during the procedure at three-minute intervals until the removal of the isolation system.
  Five minutes after the participant is seated on the dental chair, a pulse oximeter (OxyWatch, ChoiceMMed, Hamburg, Germany) will be placed on the right forefinger to record the heart rate per minute.
Systolic and Diastolic blood pressure in millimeters of mercury (mmHg) | Baseline before starting the dental procedure and then during the procedure at three-minute intervals until the removal of the isolation system.
  Five minutes after the participant is seated on the dental chair, an automatic blood pressure cuff will be applied to the left upper to record the blood pressure in millimeters of mercury (mmHg).
Behavioral pain and discomfort | During the dental procedure
  The dental procedure will be videotaped using a high-resolution camera fixed in the clinic. The recorded videos will be used to assess the participants' behavioral pain and discomfort using the Face, Legs, Activity, Cry, Consolability (FLACC) scale two trained and calibrated evaluators independently.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Bagher, Mater, Principal Investigator — Associate Professor
Locations (1):
- King AbdulAziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No